CLINICAL TRIAL: NCT00848458
Title: Azelaic Acid Iontophoresis Versus Topical Azelaic Acid Cream in the Treatment of Melasma - An Open Randomized, Controlled, Prospective, Single Blinded Clinical Trial
Brief Title: Azelaic Acid Iontophoresis Versus Topical Azelaic Acid Cream in the Treatment of Melasma
Acronym: AAI
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Schmidt.JB.MD, Department of Dermatology / MUV
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAI; Eudra-CT Number:2008-003792-52
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2010-07-15 (Estimated); Status verified 2010-07

CONDITIONS: Melasma
Keywords: Azelaic Acid; Iontophoresis
MeSH Terms: conditions — Melanosis | interventions — Iontophoresis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Azelaic Acid Iontophoresis (Experimental)
  Interventions: Other: Iontophoresis
- Azelaic acid topical (Active Comparator)
  Interventions: Other: Azelaic acid cream

INTERVENTIONS:
Other: Iontophoresis — iontophoresis with 15% azelaic acid gel twice weekly
  Arms: Azelaic Acid Iontophoresis
Other: Azelaic acid cream — topical treatment with 20% azelaic acid cream twice daily
  Arms: Azelaic acid topical

SUMMARY:
The purpose of this prospective, randomized, controlled, single-blinded investigation is to study the efficacy, tolerability and safety of azelaic acid iontophoresis (AAI) versus topical treatment with azelaic acid cream in female patients with melasma.

DETAILED DESCRIPTION:
Patients will be randomized and allocated in concealed manner to one of the two treatment arms: AAI or topical azelaic acid cream.

Azelaic acid iontophoresis treatment schedule:

Patients randomized to the AAI group will receive iontophoresis with 15% azelaic acid twice weekly over a period of 12 weeks.

Azelaic acid topical treatment schedule:

Patients randomized to the topical treatment group will receive topical treatment with 20% azelaic acid cream twice daily over a period of 12 weeks.

Besides emollients no additional specific treatments will be allowed during the study.

The use of broad spectrum (UVA+UVB) sunscreen is recommended over the entire study period (9 month).

Follow-up period:

After completion of the active study period (3 month in both treatment groups), maintenance and efficacy of both treatment schedules will be followed up quarterly over 6 month

ELIGIBILITY:
Inclusion Criteria:

* Woman
* MASI - Score over 6
* Age: over 18 years
* Skin Type: III, IV, V

Exclusion Criteria:

* Skin Type: I, II, VI
* Pregnant or lactating women
* Local therapy of intent-to-treat area within the last 6 month
* Patient with a pacemaker or metal implant
* Epileptic
* Mental incompetence to understand the protocol
* Known allergic reactions to one of used substances
* Serious encroachment on physical condition

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Change in colorimetric measurement of skin colour and MASI-Score after 12 weeks of treatment | 3 month

SECONDARY OUTCOMES:
Physician Global Assessment, Patient Global Assessment, Overall Response Assessment | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: JB Schmidt, MD, Principal Investigator — MUV; Oliver Schanab, MD, Study Director — MUV
Locations (1):
- Medical University Vienna / Depatment of Dermatology, Vienna, Austria